CLINICAL TRIAL: NCT06763367
Title: Clinical Evaluation and Study of the Efficacy of a Centella Asiatica-Infused Facial Mask on Discosmetic Dermatosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, dai jie, Nanjing First Hospital, Nanjing Medical University., Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20241217-04
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Rosacea; Acne; Centella; Melasma
MeSH Terms: conditions — Rosacea; Acne Vulgaris; Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Containing Centella sinensis mask group (Experimental): According to the random number table, both sides of the subjects' faces were randomly divided into the mask side and the control side (made of the same mask-like dressing), that is, one side of the face was applied with the Besuquan moisturizing repair mask, and the other side was applied with the control side. Patients were followed up on the day of treatment and 1, 2, 3, 4, 6 and 8 weeks after treatment. The specific methods are as follows: The patient applied 3 lobed membranes per week for the first month, and 2 pieces per week for 20 minutes each time for the second month.
  Interventions: Other: Face mask containing Centella sinensis

INTERVENTIONS:
Other: Face mask containing Centella sinensis — A half-face control test was used in this study. One side of the face was treated with a mask containing Asiaticum asiatica and the other side was treated with a mask without Asiaticum asiatica

SUMMARY:
The purpose of this study was to investigate the efficacy and safety of repairing facial mask containing Asiaticum asiatica in treating disjunctive skin diseases. A multi-center randomized double-blind self-half face control method was used. A computer-generated randomization method was used. Each cheek was randomly assigned to receive the snow glycoside mask and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Meet mild to moderate rosacea, acne diagnostic criteria; Meet the diagnostic criteria for melasma;
2. Over 18 years of age;
3. Be able to follow the treatment rules of the study and be followed for 8 weeks;
4. Informed consent; 5There were no significant cardiac, liver, kidney, gastrointestinal, neurological, psychiatric, or metabolic disorders

6.No medication was used within 1 month

Exclusion Criteria:

1. Currently pregnant, planning to become pregnant or breastfeeding;
2. Documented hypersensitivity to any active ingredient or excipient included in the study drug, or a history of adverse reactions to cosmetic products;
3. Participate in other clinical studies within 3 months before the start of the study;
4. Frequent use of Chinese medicine, sleeping pills, sedatives, anti-anxiety drugs or potentially addictive substances;
5. Present with concomitant skin conditions that may confuse the clinical assessment of rosacea, melasma, seborrheic dermatitis or pose a risk to participants, or have a history of severe skin conditions;
6. Normal use of relevant treatment (including intense pulsed light, pulsed fuel laser, oral and topical tranexamic acid, oral tetracycline antibiotics, oral compound glycyrrhizin and other anti-inflammatory drugs)
7. Patients with incomplete observation data, incomplete course of treatment and inability to take drugs as prescribed by doctors were removed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-08 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical erythema Score (CEA) | Patients were followed up on the day of treatment and at 1, 2, 3, 4, 6, and 8 weeks after treatment.
  Clinical erythema score (CEA) was divided into no, mild, moderate and severe according to the severity of rosacea, corresponding to 0,1,2,3, respectively.
Global Aesthetic Improvement Scale Score (GAIS) | Patients were followed up on the day of treatment and at 1, 2, 3, 4, 6, and 8 weeks after treatment.
  The Global Aesthetic Improvement Scale (GAIS) score was evaluated by the treating physician and divided into four levels: very improved corresponding, substantial improvement, improvement, no change; Corresponding to the best beauty effect, significant improvement but not the best, significant improvement, no change;
Melasma Area and Severity Rating (MASI) | Patients were followed up on the day of treatment and at 1, 2, 3, 4, 6, and 8 weeks after treatment.
  The melasma Area and Severity Rating (MASI) is used to evaluate the severity of melasma. Melanin deposition was quantitatively evaluated from three aspects: area, color depth and color uniformity. Area weight: Forehead 30%, left cheek 30%, right cheek 30%, mandibular 10%, color plaque proportion (A) < 10% recorded 1 points, 10% ~ 29% recorded 2 points, 30% ~ 49% recorded 3 points, 50% ~ 69% recorded 4 points, 70% ~ 89% recorded 5 points, 90% ~ 100% recorded 6 points; Color depth (D), color uniformity (H) scores range from 0 to 4 points, no score 0 points, slight score 1 points, moderate score 2 points, obvious score 3 points, maximum score 4 points. MASI score = forehead [0.3A (D+H)]+ right cheek [0.3A (D+H)]+ left cheek [0.3A (D+H)]+ mandibular [0.1A (D+H)], score range 0 ~ 48, score was positively correlated with melanin deposition.

SECONDARY OUTCOMES:
Dermatology Quality of Life Score (DLQI) | Patients were followed up on the day of treatment and at 1, 2, 3, 4, 6, and 8 weeks after treatment.
  The Dermatology Life Quality Score (DLQI) is scored by answering multiple questions in which patients self-rate the impact of their current illness on their lives over a period of one week. The answer is divided into four levels, very serious 3 points, severe 2 points, a little 1 point, no 0 points; '

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided